CLINICAL TRIAL: NCT01990664
Title: A Multi-Center Clinical Evaluation of Lapsed Contact Lens Wearers Who Are Re-Fit Into Spherical or Toric Senofilcon A Contact Lenses
Brief Title: Clinical Evaluation of Lapsed Contact Lens Wearers Who Are Re-fit Into Senofilcon A Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR-5464
Record Dates: First submitted 2013-11-15; First posted 2013-11-21 (Estimated); Results first posted 2016-02-25 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2016-01

CONDITIONS: Lapsed Contact Lens Wear

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- senofilcon A (Experimental): Contact lenses to be worn in a daily wear modality
  Interventions: Device: senofilcon A
- senofilcon A for Astigmatism (Experimental): Contact lenses to be worn in a daily wear modality
  Interventions: Device: senofilcon A for Astigmatism

INTERVENTIONS:
Device: senofilcon A
  Arms: senofilcon A
Device: senofilcon A for Astigmatism
  Arms: senofilcon A for Astigmatism

SUMMARY:
This study is an open-label, multi-site study. The total number of subjects was 200. The duration of this study was approximately four weeks. The primary objective was to assess what percentage of lapsed contact wearers, who have discontinued use of their contact lenses for greater than six months can be successfully re-fit with senofilcon A, reusable 2-weekly replacement daily wear lenses (spherical and toric designs).

ELIGIBILITY:
Inclusion Criteria:

1. The subject must read, understand , and sign the Statement of Informed Consent and receive a fully executed copy of the form.
2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. The subject must be interested in wearing contact lenses.
4. The subject must be at least 18 years old or less than 40 years of age at the time of consent.
5. The subject's vertexed spherical cylindrical refraction must result in a contact lens prescription for each eye that is available in the investigator's choice of study contact lens material(s).
6. The subject must have best corrected visual acuity of 20/30 or better in each eye.
7. The subject must require visual correction in both eyes.
8. The subject must be a lapsed wearer (defined as, any non-contact lens wearer requiring optical correction who has been previously fitted in and has previously purchased contact lenses but has since discontinued contact lens wear for any reason more than 6 months prior to the time of consent).
9. The subject must have normal eyes (i.e., no ocular medications or infections of any type).

Exclusion Criteria:

1. Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued).
2. Any ocular or systemic allergies or diseases that may interfere with contact lens wear.
3. Any systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear.
4. Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or moderate or above corneal distortion.
5. Any previous, or planned, ocular or intraocular surgery (e.g., radial keratotomy, photorefractive keratectomy (PRK), LASIK, etc.)
6. Any grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA classification scale, any previous history or signs of a contact lens related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality tha may contraindicate contact lens wear.
7. Any ocular infection.
8. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
9. Participation in any contact lens or lens care trial within one year prior to study enrollment.
10. History of binocular vision abnormality or strabismus.
11. Any infectious disease (e.g., hepatitis, tuberculosis) or contagious immunosuppressive disease (e.g., HIV), by self report.
12. Employee of the investigational clinic (i.e., Investigator, Coordinator, or Technician).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 199 (Actual)
Dates: Start 2013-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Jacksonville, Florida
  - Saint Augustine, Florida
  - Sarasota, Florida
  - Roswell, Georgia
  - Bloomington, Illinois
  - Raytown, Missouri
  - Vestal, New York
  - Raleigh, North Carolina
  - Warwick, Rhode Island
  - Memphis, Tennessee

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 199 subjects were enrolled in the study; 7 subjects were enrolled but not randomized. 18 subjects were discontinued and 174 subjects completed the study. Of those 174 completed subjects, 5 subjects had major protocol deviations; 169 subjects were included in the analysis.
Groups:
- Control (Senfilcon A): Subjects that were randomized to receive the Control lens for the duration of the study.
- Test (Senofilcon A): Subjects that were randomized to receive theTest lens for the duration of the study.
Period: Overall Study
Arm/Group | Control (Senfilcon A) | Test (Senofilcon A)
Started | 102 | 90
Completed | 95 | 79
Not Completed | 7 | 11
Not completed — Lost to Follow-up | 2 | 6
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Protocol Violation | 1 | 0
Not completed — Lens Discomfort | 1 | 1
Not completed — Lens Handling Difficulties | 1 | 0
Not completed — Unsatisfactory Visual Response | 0 | 1

BASELINE CHARACTERISTICS:
Population: The analysis population consists of all subjects that were enrolled into the study
Groups:
- Control (Senfilcon A): Consists of subjects that were dispensed at least one Control lens.
- Test (Senofilcon A): Consists of subjects that were dispensed at least one Test lens.
- Total: Total of all reporting groups
Arm/Group | Control (Senfilcon A) | Test (Senofilcon A) | Total
Number analyzed (Participants) | 102 | 90 | 192
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.80 (6.356) | 29.22 (5.715) | 29.57 (6.096)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 62 | 131
  Male | 33 | 28 | 61
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Black or African American | 20 | 22 | 42
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  White | 78 | 65 | 143
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 102 | 90 | 192

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Successfully Re-fitted Subjects
Description: Percentage of lapsed contact wearers who were successfully refitted among subjects who have lapsed from contact lens use more than 6 months prior to the date of enrollment in the study. Successful fit was assessed by on eye care practitioner (ECP) judgment of acceptable physiology.
Time Frame: 4 weeks
Population: The analysis population includes all subjects who have completed all study visits without a major protocol deviation.
Measure: Number; unit: percentage of Subjects
Groups:
- Control (Senofilcon A): Subjects that were randomized to receive the Control lens for the duration of the study.
- Test (Senofilcon A): Subjects that were randomized to receive the Test lens for the duration of the study.
Arm/Group | Control (Senofilcon A) | Test (Senofilcon A)
Number analyzed (Participants) | 93 | 76
percentage of Subjects | 100 | 95.52

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study- approximately 5 months
Arm/Group | Control (Senofilcon A) | Test (Senofilcon A)
Serious Adverse Events (participants affected / at risk) | 0/102 | 0/90
Other Adverse Events (participants affected / at risk) | 0/102 | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days